CLINICAL TRIAL: NCT04537988
Title: ECHANGE: Using EHealth Design to Facilitate Weight Maintenance Following Initial Weight Loss
Brief Title: ECHANGE: EHealth Design to Facilitate Weight Maintenance Following Initial Weight Loss
Acronym: eCHANGE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Sorlandet Hospital HF (Other Government); University of Twente (Other); Mayo Clinic (Other); The Hospital of Vestfold (Other)
Responsible Party: Principal Investigator, Lise Solberg Nes, Head of Department, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20/13923
Record Dates: First submitted 2020-06-24; First posted 2020-09-03 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Weight, Body
Keywords: Weight maintenance
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Intervention Model Description: Testing a prototype of an eHealt self-management intervention of long-term weight loss maintenance to evaluate usability and preliminary efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Feasibility and usability intervention trial (Experimental): Pre-post evaluation of a 3-month pilot-trial of an electronic health (eHealth) intervention
  Interventions: Other: Behavioral: eCHANGE

INTERVENTIONS:
Other: Behavioral: eCHANGE — eCHANGE is an eHealth intervention aiming to support long-term weight maintenance after initial weight loss

SUMMARY:
The aim of this study is to evaluate an eHealth intervention facilitating weight maintenance following initial weight loss during a 3-month trial (pilot test)

DETAILED DESCRIPTION:
Obesity rates are rapidly increasing and even with diets and interventions aiding weight loss, an alarmingly large percentage of people struggle to maintain the lost weight. In the face of obesity, weight maintenance is therefore arising as a major obstacle and new innovative approaches are called for. Despite the fact that a substantial number of web-based diets, health and fitness focused interventions or "apps" already exist, few focus on weight maintenance, are research based or available post study. In addition, most have yet to show short- or long-term effect and few, if any, are developed together with users (e.g., patients, health care professionals). eHealth solutions may therefore be a "missing link" in supporting self-regulation and motivation for sustainable health behavior change and weight loss maintenance. The aim of this study is to evaluate a person-centered, evidence based interactive eHealth intervention facilitating weight maintenance following initial weight loss during a 3- month feasibility pilot trial.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30 or more before weight loss
* 8% weight reduction or more through conservative methods
* Aim to maintain weight after weight loss or prevent weight gain
* Understand and read the Norwegian languague
* Can access the internet and own a smartphone

Exclusion Criteria:

* Weight loss through surgery or medication
* Medication to support weight loss or maintenance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy and usability | Baseline and at 3 months post baseline
  Collected data from system use log and from study specific system usefulness questions (use and perceived usefulness)

SECONDARY OUTCOMES:
Weight | Baseline and at 3 months post baseline
  Weight measurement

OTHER OUTCOMES:
Three-Factor Eating Questionnaire (TFEQ-R21) | Baseline and at 3 months post baseline
  21 item scale to evaluate cognitive restraint, emotional eating and bingeing behaviors
Pittsburgh Sleep Quality Index (PSQI) | Baseline and at 3 months post baseline
  A self-reporting questionnaire of 19 individual items, creating 7 components that produce one global score.
System Usability Scale (SUS) | At 3 months post baseline
  1o item scale measuring usability, with five response options for respondents; from Strongly agree to Strongly disagree. The obtainable score range is 25 to 100. A SUS score above a 68 would be considered above average and anything below 68 is below average.
TWente Engagement with Ehealth Technologies Scale (TWEETS) | At 3 months post baseline
  To measure behavioral, cognitive and affective engagment with a 5 point Likert scale: strongly disagree, disagree, neutral, agree, strongly agree
The Hospital Anxiety and Depression Scale (HADS) - Assessing change | At baseline and at 3 months post baseline
  14 item scale measuring anxiety and depression. Respondents are asked to indicate which of 4 response options (rated from 0-3; score range, 0-42) comes closest to describing how they have been feeling in the previous week for each item. Scores from 0-7 on the subscales are regarded as being in the normal range; a score of 11 or higher indicates a probable presence of a mood disorder, and a score of 8-10 is suggestive of the presence of the state.
RAND Health Related Quality of Life | 36 item scale measuring health related quality of life. The RAND-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question
  At baseline and at 3 months post baseline
Weight-related Symptom Measure (WRSM) | At baseline and at 3 months post baseline
  Patient reported outcome measures that assesses the symptoms that are commonly associated with obesity, next to quality of life, general functional status and well-being.
Treatment Self-Regulation Questionnaire (TSRQ diet and exercise) | At baseline and at 3 months post baseline
  A theoretically derived scale which assesses the degree of autonomous self-regulation regarding why people engage or would engage in healthy behavior
Perceived Competence Scale (PCS) (diet and exercise) | At baseline and at 3 months post baseline
  A 4-item questionnaire, that assesses participants' feelings of competence about engaging in a healthier behavior (e.g., diet) and participating in a physical activity regularly.

CONTACTS AND LOCATIONS:
Overall Officials: Lise Solberg Nes, PhD, Principal Investigator — Head of Department
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Asbjornsen RA, Hjelmesaeth J, Smedsrod ML, Wentzel J, Ollivier M, Clark MM, van Gemert-Pijnen JEWC, Solberg Nes L. Combining Persuasive System Design Principles and Behavior Change Techniques in Digital Interventions Supporting Long-term Weight Loss Maintenance: Design and Development of eCHANGE. JMIR Hum Factors. 2022 May 27;9(2):e37372. doi: 10.2196/37372. PMID 35622394
- [Derived] Asbjornsen RA, Wentzel J, Smedsrod ML, Hjelmesaeth J, Clark MM, Solberg Nes L, Van Gemert-Pijnen JEWC. Identifying Persuasive Design Principles and Behavior Change Techniques Supporting End User Values and Needs in eHealth Interventions for Long-Term Weight Loss Maintenance: Qualitative Study. J Med Internet Res. 2020 Nov 30;22(11):e22598. doi: 10.2196/22598. PMID 33252347